CLINICAL TRIAL: NCT00005319
Title: Epidemiologic Studies of Blood Use in the United States - SCOR in Transfusion Medicine
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4093; P50HL033774 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2002-05

CONDITIONS: Blood Transfusion

SUMMARY:
To develop and apply quantitative methods by which to measure and characterize blood transfusion practice in specific diagnoses and procedures; to open scientific communication about transfusion practice within and across institutions; and to develop simpler methods for estimating annual national blood collections and transfusions.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The study was a subproject within a Specialized Centers of Research (SCOR) in Transfusion Medicine. The experimental design was based on the study and analysis of several unique sets of data. One set consisted of abstracted patient data including ICD-9-CM diagnosis and procedure, DRG and red cell units transfused, from a constant set 100 of United States hospitals for the years 1980,82,84,86, to which a new set of data was added for the year 1989. A similar set of data were gathered from eight cooperating teaching hospitals over the first four years of the grant term; this set included data for transfusions of all blood components, autologous units and factor preparations. A third data base contained the data for four United States surveys conducted in 1982,84,86,87; and was expanded to include 1990 and 92. Using these data, four main tasks were addressed. A Pan-DRG red cell transfusion study was conducted to ascertain red cell use across all DRGs and ICD-9-CM codes. Extensive efforts were devoted to developing new methods to characterize transfusion practice. A series of studies were devoted to characterizing transfusions of all blood components in a selected number of ICD-9-CM classes. The purpose of the fourth task was to develop simpler and more rapid alternative methods for producing national estimates of transfusion activity; as part of this task,new surveys were conducted for 1990 and 92.

Among the questions studied were: Was it possible to identify distinctive attributes of the patients who, though operated, did not require a transfusion or who required a large volume of blood? Were transfusions of non-red cell components related to use of red cells? Could transfusion frequency diagnosis for all blood products be used as a measure of transfusion practice? Did longitudinal comparisons of transfusions over the 9-year interval, 1980-1989, reveal significant trends? Was it possible to discriminate quantitatively between transfusion practices in different hospitals or set of hospitals, or at different times? What was the effect of autologous blood programs in transfusion practice? What was the contribution of comorbid conditions on red cell and component transfusion patterns.?

The dollars for the subproject were approximately 25 percent of total dollars spent each year for the Center.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 1996-12 (Actual)

REFERENCES:
- [Background] Wallace EL, Churchill WH, Surgenor DM, Cho GS, McGurk S. Collection and transfusion of blood and blood components in the United States, 1994. Transfusion. 1998 Jul;38(7):625-36. doi: 10.1046/j.1537-2995.1998.38798346630.x. PMID 9683100
- [Background] Churchill WH, McGurk S, Chapman RH, Wallace EL, Bertholf MF, Goodnough LT, Kao KJ, Olson JD, Woodson RD, Surgenor DM. The Collaborative Hospital Transfusion Study: variations in use of autologous blood account for hospital differences in red cell use during primary hip and knee surgery. Transfusion. 1998 Jun;38(6):530-9. doi: 10.1046/j.1537-2995.1998.38698326332.x. PMID 9661686
- [Background] Surgenor DM, Churchill WH, Wallace EL, Rizzo RJ, McGurk S, Goodnough LT, Kao KJ, Koerner TA, Olson JD, Woodson RD. The specific hospital significantly affects red cell and component transfusion practice in coronary artery bypass graft surgery: a study of five hospitals. Transfusion. 1998 Feb;38(2):122-34. doi: 10.1046/j.1537-2995.1998.38298193094.x. PMID 9531943
- [Background] Wallace EL, Churchill WH, Surgenor DM, An J, Cho G, McGurk S, Murphy L. Collection and transfusion of blood and blood components in the United States, 1992. Transfusion. 1995 Oct;35(10):802-12. doi: 10.1046/j.1537-2995.1995.351096026360.x. PMID 7570909
- [Background] Churchill WH, Chapman RH, Rutherford CJ, Poss R, Wallace EL, Surgenor DM. Blood product utilization in hip and knee arthroplasty: effect of gender and autologous blood on transfusion practice. Vox Sang. 1994;66(3):182-7. doi: 10.1111/j.1423-0410.1994.tb00307.x. PMID 8036787
- [Background] Wallace EL, Surgenor DM, Hao HS, An J, Chapman RH, Churchill WH. Collection and transfusion of blood and blood components in the United States, 1989. Transfusion. 1993 Feb;33(2):139-44. doi: 10.1046/j.1537-2995.1993.33293158046.x. PMID 8430453
- [Background] Surgenor DM, Wallace EL, Churchill WH, Hao SH, Chapman RH, Collins JJ Jr. Red cell transfusions in coronary artery bypass surgery (DRGs 106 and 107). Transfusion. 1992 Jun;32(5):458-64. doi: 10.1046/j.1537-2995.1992.32592327721.x. PMID 1626350
- [Background] Surgenor DM, Wallace EL, Churchill WH, Hao SH, Chapman RH, Poss R. Red cell transfusions in total knee and total hip replacement surgery. Transfusion. 1991 Jul-Aug;31(6):531-7. doi: 10.1046/j.1537-2995.1991.31691306252.x. PMID 1906649
- [Background] Surgenor DM, Wallace EL, Hao SH, Chapman RH. Collection and transfusion of blood in the United States, 1982-1988. N Engl J Med. 1990 Jun 7;322(23):1646-51. doi: 10.1056/NEJM199006073222306. PMID 2342524
- [Background] Surgenor DM, Wallace EL, Churchill WH, Hao S, Hale WB, Schnitzer J. Utility of DRG and ICD-9-CM classification codes for the study of transfusion issues. Transfusions in patients with digestive diseases. Transfusion. 1989 Nov-Dec;29(9):761-7. doi: 10.1046/j.1537-2995.1989.29990070178.x. PMID 2686107
- [Background] Surgenor DM, Wallace EL, Hale SG, Gilpatrick MW. Changing patterns of blood transfusions in four sets of United States hospitals, 1980 to 1985. Transfusion. 1988 Nov-Dec;28(6):513-8. doi: 10.1046/j.1537-2995.1988.28689059022.x. PMID 3194926
- [Background] Surgenor DM, Churchill WH, Wallace EL, Rizzo RJ, Chapman RH, McGurk S, Bertholf MF, Goodnough LT, Kao KJ, Koerner TA, Olson JD, Woodson RD. Determinants of red cell, platelet, plasma, and cryoprecipitate transfusions during coronary artery bypass graft surgery: the Collaborative Hospital Transfusion Study. Transfusion. 1996 Jun;36(6):521-32. doi: 10.1046/j.1537-2995.1996.36696269511.x. PMID 8669084